CLINICAL TRIAL: NCT04038125
Title: Increase in Capillary Plexus Density Level Following the Use of Ozurdex for the Treatment of DME (RMSM ICOD STUDY)
Brief Title: Increase in Capillary Plexus Density Level Following the Use of Ozurdex for the Treatment of DME
Acronym: ICOD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Retina Macula Specialists of Miami, LLC (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Diana Shechtman, OD FAAO, Principal Investigator - OD, FAAO, Retina Macula Specialists of Miami, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCH-0-012-019
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy; Retinal Ischemia
Keywords: Diabetic Macula Edema; Diabetic Retinopathy; Retina Ischemia
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ozurdex Implant (Other): Intravitreal injection of Ozurdex implant
  Interventions: Drug: Ozurdex Drug Implant Product

INTERVENTIONS:
Drug: Ozurdex Drug Implant Product — Intravitreal Ozurdex injection
  Other Names: Dexamethasone

SUMMARY:
The objective of this study is to test the hypothesis that following the use of intravitreal dexamethasone implant for the treatment of DME, there will be an observable increase in the capillary density plexus as denoted by the quantitative assessment of the superficial capillary plexus on OCTA, as well as a decrease in size of the foveal avascular zone (FAZ).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and Older.
2. Diagnosis of diabetes mellitus (type 1 or type 2).
3. At least one eye meets the study eye criteria listed.
4. Visual Acuity 20/30 - 20/200 Snellen equivalent
5. Have received no previous treatment for diabetic macular edema,(treatment naïve)
6. Mild to Severe Non-proliferative Diabetic Retinopathy
7. Diabetic macular edema present on optical coherence tomography (OCT) central subfield: ≥ 300µm.
8. Able and willing to provide informed consent.

Exclusion Criteria:

1. Have had any prior ocular treatment.
2. Have had prior retinal surgical ( i.e. Pars plana vitrectomy). 3 .Have any clinical evidence of proliferative diabetic retinopathy.

4. Have a HBA1c of greater of 10%. 5. Evidence of Glaucoma or who are labeled glaucoma suspect at screening (defined as C/D >/= 0.5 with correlated NFLA thinning or IOP>25mmHg). 6. Have a contraindication to Ozurdex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate re perfusion following Ozurdex use. | 6 Months
  Determined by OCT-A

CONTACTS AND LOCATIONS:
Overall Officials: Diana Shechtman, OD FAAO, Principal Investigator — Retina Macula Specialists of Miami, LLC
Locations (2):
- United States (2):
  - Retina Macula Specialists of Miami, LLC, North Miami Beach, Florida
  - Retina Macula Specialists of Miami, LLC, South Miami, Florida